CLINICAL TRIAL: NCT07397715
Title: Association of Ultrasound Features of the Myometrium Suggestive of Adenomyosis and Clinical Symptoms (MUSA 3)
Brief Title: Association of Ultrasound Features of the Myometrium Suggestive of Adenomyosis and Clinical Symptoms
Acronym: MUSA3
Status: Recruiting | Type: Observational
Sponsor: Swiss GO Trial Group (Network)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Swiss-GO-09/BASEC:2023-01484; 2023-01484 (Other: Swissethics)
Record Dates: First submitted 2025-05-13; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Adenomyosis of Uterus
Keywords: Adenomyoma; Deep infiltrating endometriosis; Gynaecological transvaginal ultrasound; Gynaecological Ultrasound; Myometrium; Uterine anomaly; Asymptomatic adenomyosis; Symptomatic adenomyosis; Menstrual bleeding; Bleeding disorders; Abnormal uterine bleeding; Abdominal pain; Dysmenorrhoea; Dyspareunia; Morphological Uterus Sonographic Assessment (MUSA); Adenomyosis Grading; Subfertility; Ultrasound features; Myometrial cysts; Hyperechogenic island; Echogenic subendometrial lines and buds; Globular uterus; Asymmetrical myometrial thickening; Fan shaped shadowing; Cyclical/non-cyclical bleeding; menorrhagia; Metrorrhagia; Translesional vascularity; Irregular junctional zone; Interrupted junctional zone; benign fibroid; Myoma
MeSH Terms: conditions — Adenomyosis; Adenomyoma; Uterine Anomalies; Hemostatic Disorders; Metrorrhagia; Abdominal Pain; Dysmenorrhea; Dyspareunia; Infertility; Menorrhagia; Myoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with a uterus: Pre - and perimenopausal women with a uterus that are scheduled for a gynaecologic ultrasound exam.

SUMMARY:
The goal of this study/research is to assess the relationship between ultrasound features of the myometrium suggestive of adenomyosis and clinical symptoms of adenomyosis and to establish a reporting system for adenomyosis assessing disease severity. Consecutive pre- and perimenopausal symptomatic and asymptomicasymptomatic women with an uterus presenting for gynaecological ultrasound exams will be asked to participate in the study. Routine gynecologicalgynaecological ultrasound exams will be performed and study participants will fill out a questionnaire on their symptoms (if any) and bleeding pattern. There will be one visit and no interventions.

DETAILED DESCRIPTION:
In adenomyosis endometrial tissue is embedded in the myometrium of the uterus. It is considered a relevant benign, underreported disease of the uterus and is a frequent cause of dysmenorrhea, bleeding disorders and abdominal pain and subfertility. The reference standard for diagnosis is histology, but the majority of women will have hormonal medical treatment, are in the reproductive age and will not undergo surgery (i.e. hysterectomy). Today ultrasound has become the first line imaging method for diagnosis.

The proportion of women that show ultrasound features of adenomyosis without symptoms is unknown but a third of young, nulliparous women without other associated disease will show signs of adenomyosis.

The MUSA consensus describes ultrasound features suggestive of adenomyosis: asymmetrical thickening of the myometrium, cysts within the myometrium, echogenic subendometrial lines and buds, hyperechoic islands, fan shaped shadowing and an irregular or interrupted junctional zone. More recently the MUSA criteria have been specified further and now distinguish between direct features, that are typical for adenomyosis and indirect features that result from ectopic endometrium in the myometrium.

This is a cross sectional exploratory non-interventional observational multicenter study with one visit and no interventions with assessment of participant demographics, standardized assessment of bleeding, standardized assessment of pain, standardized ultrasound exam.

The primary objective of the study is to assess the relationship between MUSA-defined ultrasound features of the myometrium suggestive of adenomyosis and the severity of clinical symptoms, specifically pain (NRS) and abnormal uterine bleeding (PBAC).

Secondary objectives are:

* to identify which individual ultrasound features best explain variation in symptom severity scores.
* to estimate the prevalence of ultrasound features in different subgroups of women, including symptomatic and asymptomatic participants.
* to develop an exploratory ultrasound-based grading system for adenomyosis that integrates MUSA features with clinical symptom severity.

The participants are consecutively enrolled at the sites when they present for a scheduled gynecologic ultrasound exam, fit the inclusion criteria, and do not have any positive exclusion criteria.

The files or referrals of the participants will be screened for eligibility at the participating site's department. Participants will be included if they have signed the consent for the study (ideally prior to the ultrasound exam, but recruitment after the routine exam is also possible). Since the ultrasound data is assessed within routine care the additional exam time for the participants should be almost unchanged. The filling out of the questionnaire for assessment of pain and bleeding will take some extra time (10-15min). The clinical and ultrasound data will be entered into the electronic patient file immediately by the examiner and the transfer into the data miner will occur within one month of the ultrasound exam by the examining physician or a member of the study team.

The investigators plan to include 1000 participants from at least seven centres in Europe and Switzerland. Out of that the investigators plan to include 400 from Switzerland. The study duration is estimated to be three years.

ELIGIBILITY:
Inclusion Criteria:

* Women of pre- and perimenopausal age presenting for gynaecologic ultrasound exam giving voluntary informed written consent.
* Symptomatic and asymptomatic women
* Patients with hormonal contraceptives and Hormone Replacement Therapy (HRT) can be included, but information will be noted.

Exclusion Criteria:

* Missing written consent (study consent)
* Any serious underlying medical, psychiatric or psychological condition, which may interfere with the patient's capacity of discernment.
* Postmenopausal women
* Pregnancy
* History of pelvic urogynaecologic surgery (TVT, mesh surgery, etc.)
* Malignancy or premalignancy of uterus/cervix
* Prior myomectomy for FIGO 3-6 fibroids
* Patients with coagulation disorders under current anticoagulation medication
* Prior history of diagnosed intraabdominal adhesions (surgery)
* Prior diagnosis of pelvic congestion syndrome
* Psychiatric disease precluding a reliable estimation of pain
* Prior surgery or treatment for deep infiltrating endometriosis
* Acute other symptoms:
* Urinary symptoms (dysuria, urgency, grade III stress incontinence)
* Acute of chronic pelvic infection (cervicitis, endometritis, salpingitis, frozen pelvis)
* Ovarian lesions
* Sonographic signs of deep infiltrating endometriosis (DIE)
* Intracavitary pathology (Fibroid 0-2, polyp, adhesions)
* Retained products of conception
* >3 small fibroids below 2 cm in largest diameter FIGO 3-8 (i.e. the presence of three fibroids below 2cm is NOT considered an exclusion criterion)
* Presence of any fibroid >2cm.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women of pre- and perimenopausal age presenting for gynaecologic ultrasound exam giving voluntary informed written consent.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Association between MUSA defined ultrasound features of adenomyosis and the severity of clinical symptoms. | At baseline (single assessment at the time of the routine ultrasound examination)
  The correlation between the total number of MUSA defined ultrasound features (presence/absence; feature count) and clinical symptom severity will be assessed using the Numeric Rating Scale (NRS 0-10) for pain and the Pictorial Blood Assessment Chart (PBAC) score for abnormal bleeding. The primary outcome will be expressed as a correlation coefficient (unitless).

SECONDARY OUTCOMES:
Association of individual ultrasound features with symptom severity | At baseline (single assessment at the time of the routine ultrasound examination)
  Each individual MUSA defined ultrasound feature (binary: yes/no) will be evaluated for its association with pain severity (NRS 0-10) and bleeding severity (PBAC score). Results will be reported as an effect size or correlation coefficient (unitless).
Prevalence of individual MUSA defined features | At baseline (single assessment at the time of the routine ultrasound examination.
  The proportion of participants who exhibit each individual MUSA defined ultrasound feature will be reported.
Prevalence of Ultrasound Features in Symptomatic vs. Asymptomatic Participants | At baseline (single assessment at the time of the routine ultrasound examination
  The percentages of symptomatic participants (pain and/or abnormal bleeding) and asymptomatic participants exhibiting each MUSA defined ultrasound feature will be compared.

OTHER OUTCOMES:
Exploratory Development of an Ultrasound Based Severity Grading System | At baseline (single assessment at the time of the routine ultrasound examination).
  An exploratory grading system integrating MUSA defined ultrasound findings with clinical symptom scores (NRS and PBAC) will be developed to propose a categorical severity classification for adenomyosis.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolin Manegold-Brauer, Prof. Dr., Principal Investigator — Deputy Head Physician, Obstetrics and Prenatal Medicine
Locations (3):
- Medical University of Silesia, Sosnowiec, Poland
- Hospital Universitari Dexeus, Barcelona, Spain
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Parties can use and may share Data under their custodianship with any third party providing analyses within the Project, if and to the extent required for the Project, provided that the Data: (i) are disposed in accordance with all necessary patient consents, regulatory approvals and the purpose of the Project, under terms at least equivalent to those of this Consortium Agreement and the data transfer and use agreement(s) and (ii) remain confidential and are published only after the publication of the results from the currently planned project and after approval of the Steering Committee.
Supporting Information: ICF
Time Frame: The estimated time time from which the data will become available will be from 1st of February 2029 onwards.
Access Criteria: Access to, provision and exchange of data, including the metadata, between the Parties under the Project (Data) shall be carried out pursuant to the Data Transfer and Use Agreement by the Parties for accessing, providing or exchanging Data under the Project.